CLINICAL TRIAL: NCT05227092
Title: 3D OPTIMIZED WMN MPRAGE Increased Detection of Focal Spinal Cord Lesion in Multiple Sclerosis (WHINUME)
Acronym: WHINUME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2021/59
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: MS; MRI; CIS; RRMS; PPMS; MPRAGE
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D OPTIMIZED WMN MPRAGE (Experimental): * At the cervical level the conventional data set: 2D Sagittal T2 FSE/ 2D Sagittal STIR / 2D Sagittal PSIR / 3D MPRAGE and the 3D OPTIMIZED MPRAGE WMN data set with sagittal and axial acquisition.
  * At the thoracic level the conventional data set: 2D Sagittal T2 FSE/ 2D Sagittal STIR / 3D MPRAGE and the 3D Sagittal OPTIMIZED MPRAGE WMN data set.
  Interventions: Device: 3D OPTIMIZED WMN MPRAGE

INTERVENTIONS:
Device: 3D OPTIMIZED WMN MPRAGE — * At the cervical level the conventional data set: 2D Sagittal T2 FSE/ 2D Sagittal STIR / 2D Sagittal PSIR / 3D MPRAGE and the 3D OPTIMIZED MPRAGE WMN data set with sagittal and axial acquisition.
  * At the thoracic level the conventional data set: 2D Sagittal T2 FSE/ 2D Sagittal STIR / 3D MPRAGE and the 3D Sagittal OPTIMIZED MPRAGE WMN data set.

SUMMARY:
The aim of this study is to compare the 3D OPTIMIZED MPRAGE WMN sequence to "conventional sequences" used in spinal cord analysis.

The patients will be explored at the cervical level with the conventional 2D sagittal T2 FSE, 2D sagittal STIR, 2D sagittal PSIR, 3D T1 MPRAGE sequences, and the sequence of interest 3D sagittal OPTIMIZED WMN MPRAGE and 3D axial OPTIMIZED WMN MPRAGE. At the thoracic level, with the conventional 2D sagittal T2 FSE, 2D sagittal STIR, 3D T1 MPRAGE sequences and the sequence of interest 3D sagittal OPTIMIZED WMN MPRAGE.

DETAILED DESCRIPTION:
Multiple sclerosis is a common inflammatory disease of the central nervous system and the leading cause of non-traumatic physical disability in young adults.

Spinal cord involvement is common, affecting approximately 90% of patients, and can be revealed by sensory loss, neuropathic pain, spasticity, motor weakness, and bladder and bowel dysfunction. Spinal cord imaging plays an important role in the diagnosis of the disease, but also in the prognosis, particularly with regard to the location and severity of the damage.

Due to the location, small size and mobility of the spinal cord, its imaging raises technical problems and fewer studies have focused on spinal cord involvement in MS than on brain involvement.

Currently, the 2D sagittal T2 FSE sequence is the imaging of choice for spinal cord analysis. Numerous sequences have been developed recently, some of which show an increase in sensitivity at the cervical level, such as short tau inversion recovery (STIR) and phase sensitive inversion recovery (PSIR). The lesion load assessed on these conventional sequences lacks correlation with clinical status, probably due to a multifactorial mechanism of disability in MS, but also probably due to the limitations of the resolution of current sequences.

WHINUME study will investigate at the spinal cord level the interest of an optimised MP-RAGE sequence cancelling the spinal cord white matter signal. The hypothesis is that this sequence could have a good sensitivity, specificity and reproducibility between readers for the detection of spinal cord lesions compared to other sequences at the cervical level but also at the thoracic level. Therefore, it could replace the conventional sequences currently available.

This study will prospectively include 60 patients with multiple sclerosis confirmed by the McDonald 2017 criteria. All patients will sign a consent form. The 3D OPTIMIZED MPRAGE WMN will be compared to conventional sequences.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* CIS or RRMS
* Medullary symptomatology less than 6 months
* With or without an objective lesion on a subsequent MRI scan
* Signed the Informed Consent

Exclusion Criteria:

* Pregnant or potentially pregnant women
* Breastfeeding woman
* Contraindications to MRI
* Other diagnosis (Neuro-myelitis spectrum disease or Progressive Multiple Sclerosis)
* Surgical history on the spinal cord or lumbar spine
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
lesions at the cervical level | day 1
  number of lesions at the cervical level for the 3D optimized WMN MPRAGE sequence compared to "conventional sequences"

SECONDARY OUTCOMES:
lesions at the thoracic level | day 1
  The number of lesions at the thoracic level for the 3D optimized WMN MPRAGE sequence compared to "conventional sequences"
sensitivity of the 3D optimised WMN MPRAGE sequence | day 1
  For the total number of lesions detected, the sensitivity of the 3D optimised WMN MPRAGE sequence compared to "conventional sequences".
positive predictive value of the 3D optimized WMN MPRAGE sequence | day 1
  For the total number of lesions detected and the positive predictive value of the 3D optimized WMN MPRAGE sequence compared to "conventional sequences
Intraclass corelation coefficient | day 1
  The reproducibility of the number of lesions will be assessed via two radiologists analysing the 3D WMN MPRAGE sequences and the "conventional sequences" twice
pathogenicity of the lesions | day 1
  Confidence in the pathogenicity of the lesions with a quantitative scale on each lesion detected at the cervical and thoracic level: 1) corresponding to a very low confidence, 2) moderate and 3) a very high confidence.
presence of artefacts | day 1
  The presence of artefacts at the cervical and thoracic level defined by a confidence scale: 1) corresponding to no artefacts, 2) minor artefacts, 3) moderate artefacts, 4) major artefacts, and 5) major artefacts
volume of lesion | day 1
  The volume (mm3) for 20 randomly selected patients, using a distinct, visible lesion at the cervical level to be detected on the "sequence of interest" and "conventional sequences".
contrast-to-noise ratio | day 1
  The contrast-to-noise ratio (CNR) calculated with [CNR = (Lesion Signal - Cord Signal) / Noise] for 20 randomly selected patients, using a distinct, visible lesion at the cervical level to be detected on the "sequence of interest" and "conventional sequences".
patient's disability | day 1
  The assessment of the patient's disability using the EDSS clinical scale (from 0-normal neurologic exam to 100-death).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No